CLINICAL TRIAL: NCT00009620
Title: Randomized Clinical Trial of Antenatal Phenobarbital in the Prevention of Neonatal Intracranial Hemorrhage
Brief Title: Antenatal Phenobarbital to Prevent Neonatal Intracranial Hemorrhage
Acronym: Phenobarbital
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Seetha Shankaran/ Lead Principal Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NICHD-NRN-0006; U10HD021385 (NIH); U10HD027881 (NIH); U10HD027871 (NIH); U01HD019897 (NIH); U10HD027856 (NIH); U10HD021415 (NIH); U10HD027880 (NIH); U10HD027853 (NIH); U10HD027851 (NIH); U10HD021364 (NIH); U10HD027904 (NIH); M01RR000997 (NIH); M01RR006022 (NIH); M01RR000750 (NIH); M01RR000070 (NIH); M01RR008084 (NIH)
Record Dates: First submitted 2001-02-01; First posted 2001-02-05 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Intracranial Hemorrhages
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Cerebral hemorrhage; Phenobarbital; Pregnancy; Prenatal care; Intraventricular hemorrhage; Periventricular leukomalacia; Brain injury; Brain hemorrhage
MeSH Terms: conditions — Premature Birth; Intracranial Hemorrhages; Cerebral Hemorrhage; Leukomalacia, Periventricular; Brain Injuries | interventions — Phenobarbital; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenobarbital (Experimental)
  Interventions: Drug: Phenobarbital
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Phenobarbital — 10 mg of phenobarbital per kilogram of body weight intravenously over a period of 20 to 40 minutes (maximal dose, 1000 mg)
  Arms: Phenobarbital
Drug: Saline — Infusion of normal sal
  Arms: Placebo

SUMMARY:
This large randomized trial tested whether phenobarbital given to a pregnant woman about to deliver a premature infant would prevent brain injuries in their newborns. Women with 24 to 32 week fetuses who were in preterm labor and were expected to deliver within 24 hrs were randomized to phenobarbital or usual care. They were treated until they deliver or the fetus reaches 33 wks gestation. Babies were followed until discharge and evaluated at 18-22 mos corrected age for neurodevelopmental outcome.

DETAILED DESCRIPTION:
The administration of phenobarbital to pregnant women before delivery has been thought to decrease the frequency of intracranial hemorrhage in preterm infants. To evaluate this potential neuroprotective therapy further, we determined the effect of antenatal administration of phenobarbital on the frequency of neonatal intracranial hemorrhage and early death. Women who were 24 to 33 weeks pregnant and who were expected to deliver their infants within 24 hours were randomly assigned to receive either intravenous phenobarbital (10 mg/kg body weight) or placebo, followed by maintenance doses until delivery or 34 wks gestation. Infants less than 34 wks at birth underwent serial cranial ultrasonography to detect the presence of intracranial hemorrhage. The sample size of 1038 pregnancies was based on an intracranial hemorrhage rate of 20 percent in the placebo and less than 12 percent in the phenobarbital group; 90 percent power; a 5 percent two-tailed type 1 error; and an 8 percent noncompliance rate. The twin with the highest grade of intracranial hemorrhage was included.

Degree of maternal sedation was evaluated after administration of study drug. Neonatal ultrasound exams were performed at 3-5 days, 10-14 days, and 38-42 wks postmenstrual age; neonatal medications were recorded during the first week of life; treatments, and outcomes were recorded through death, discharge, or 120 days, whichever occurred first. Neurodevelopmental outcome was evaluated at 18-22 months corrected age by certified examiners masked to treatment status.

ELIGIBILITY:
Inclusion Criteria:

* Admission to a high risk perinatal unit or labor and delivery unit;
* 24 to 32 completed weeks gestation;
* Expected delivery within 24 hrs;
* Preterm labor or no labor with planned delivery for maternal-fetal indications;

Exclusion Criteria:

* Anticipated delivery within two hours
* Multiple congenital or chromosomal abnormalities in the fetus
* Multiple gestation with more than two fetuses
* Administration of phenobarbital during the pregnancy
* Administration of indomethacin within one week before admission
* Maternal platelet count of less than 100,000 per cubic millimeter

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 1993-02; Primary Completion 1995-02 (Actual); Study Completion 1997-02 (Actual)

PRIMARY OUTCOMES:
Neonatal intracranial hemorrhage or death | 72 hours of life

SECONDARY OUTCOMES:
Intracranial hemorrhage (grade I, II, III, or IV) | 72 hours of life
Periventricular leukomalacia | 72 hours of life
Neurodevelopmental impairment | 18 to 22 months of corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Seetha Shankaran, MD, Study Director — Wayne State University; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Raymond Bain, PhD, Principal Investigator — George Washington University; James A. Lemons, MD, Principal Investigator — Indiana University; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee at Memphis; David K. Stevenson, MD, Principal Investigator — Stanford University; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Barbara J. Stoll, MD, Principal Investigator — Emory University; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University; William Oh, MD, Principal Investigator — Brown University, Women and Infants Hospital
Locations (11):
- United States (11):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee

REFERENCES:
- [Result] Shankaran S, Papile LA, Wright LL, Ehrenkranz RA, Mele L, Lemons JA, Korones SB, Stevenson DK, Donovan EF, Stoll BJ, Fanaroff AA, Oh W. The effect of antenatal phenobarbital therapy on neonatal intracranial hemorrhage in preterm infants. N Engl J Med. 1997 Aug 14;337(7):466-71. doi: 10.1056/NEJM199708143370705. PMID 9250849
- [Result] McCain GC, Donovan EF, Gartside P. Preterm infant behavioral and heart rate responses to antenatal phenobarbital. Res Nurs Health. 1999 Dec;22(6):461-70. doi: 10.1002/(sici)1098-240x(199912)22:63.0.co;2-t. PMID 10625862
- [Result] Shankaran S, Papile LA, Wright LL, Ehrenkranz RA, Mele L, Lemons JA, Korones SB, Stevenson DK, Donovan EF, Stoll BJ, Fanaroff AA, Oh W, Verter J. Neurodevelopmental outcome of premature infants after antenatal phenobarbital exposure. Am J Obstet Gynecol. 2002 Jul;187(1):171-7. doi: 10.1067/mob.2002.122445. PMID 12114906
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/